CLINICAL TRIAL: NCT04707703
Title: Isavuconazole for the Prevention of SARS-CoV-2-associated Invasive Aspergillosis in Critically-Ill Patients
Brief Title: Isavuconazole for the Prevention of COVID-19-associated Pulmonary Aspergillosis
Acronym: Isavu-CAPA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Participant enrollment challenges
Sponsor: Jeffrey Jenks, MD, MPH (Other)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey Jenks, MD, MPH, Assoc Physician, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 200639
Record Dates: First submitted 2021-01-08; First posted 2021-01-13 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-07

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2; Aspergillosis Invasive
Keywords: Isavuconazole; Antifungal Agents; Anti-infective Agents; Coronavirus-associated Invasive Pulmonary Aspergillosis; CAPA
MeSH Terms: interventions — isavuconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SOC plus Isavuconazonium sulfate (Experimental): SOC plus intravenous isavuconazonium sulfate 372 mg every 8 hours for 6 doses followed by 372mg once daily for up to 28 days
  Interventions: Drug: Isavuconazonium Injection [Cresemba]
- SOC plus Placebo (Placebo Comparator): SOC plus intravenous placebo every 8 hours for 6 doses followed by once daily for up to 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isavuconazonium Injection [Cresemba] — Intravenous isavuconazonium sulfate 372 mg every 8 hours for 6 doses followed by intravenous isavuconazonium sulfate 372 mg once daily for up to 28 days
  Other Names: Isavuconazole; Cresemba
  Arms: SOC plus Isavuconazonium sulfate
Drug: Placebo — Intravenous placebo every 8 hours for 6 doses followed by intravenous placebo once daily for up to 28 days
  Arms: SOC plus Placebo

SUMMARY:
The objective of this study is to evaluate whether antifungal prophylaxis with isavuconazole can reduce the incidence of SARS-CoV-2-associated invasive aspergillosis in patients in the ICU (intensive care unit) with severe COVID-19 infection.

The investigators will perform an interventional, double-blinded, randomized-controlled, multi-center study in patients with severe COVID-19 infection admitted to the ICU. Patients will be randomized to the isavuconazole prophylaxis plus standard of care (SOC) group or the placebo plus SOC group. Participants will receive isavuconazole or placebo for up to 28 days or until discharge from the hospital (whichever occurs first).

DETAILED DESCRIPTION:
Adult patients with polymerase chain reaction (PCR)-confirmed SARS-CoV-2 (COVID-19) infection without a diagnosis of invasive aspergillosis who are hospitalized in the ICU are eligible for inclusion in this study and will be randomized to the isavuconazole plus standard of care (SOC) group or placebo plus SOC group.

If randomized to the isavuconazole group, participants will receive intravenous isavuconazonium sulfate 372 mg every 8 hours for 6 doses followed by intravenous isavuconazonium sulfate 372 mg once daily for up to 28 days. If randomized to the placebo group, participants will receive intravenous placebo every 8 hours for 6 doses followed by once daily for up to 28 days. Both groups will receive the usual SOC.

Following randomized to the two treatment arms, participants will be screened for invasive aspergillosis with thrice weekly fungal cultures from tracheal aspirate (TA) secretions or thrice weekly serum galactomannan (GM) testing (if TA unable to be performed, contraindicated, or participant is not intubated). If invasive aspergillosis or other invasive fungal infection is detected, antifungal therapy will be initiated (if the participant is in the placebo arm) or modified if needed (if the participant is in the isavuconazole arm).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient or his/her legally authorized person.
* Adult patient (> 18 years).
* PCR-confirmed SARS-CoV-2 based on nasopharyngeal swab (NPS), oropharyngeal swab (OPS), tracheal aspirate (TA), bronchial aspirate (BA), or bronchoalveolar lavage fluid (BALF) within 14 days prior to ICU admission or within 72 hours following ICU admission.
* Radiographic imaging consistent with SARS-CoV-2 infection (e.g. atypical pneumonia, organizing pneumonia, ground glass opacities) or acute respiratory distress syndrome (ARDS) within 7 days of diagnosis of SARS-CoV-2 infection.
* A negative pregnancy test in women of child-bearing age.
* If a woman is of child-bearing age, she must be willing to use an effective method of contraception for 28 days after the final dose of isavuconazole per manufacturer instructions

Exclusion Criteria:

* Anticipated transfer to another medical center that is not a study site within hours of admission to the ICU.
* Pregnancy based on a positive human chorionic gonadotropin (HCG) test from serum or urine.
* Patient who is breastfeeding and unable to discontinue breastfeeding while taking the study drug.
* Patients with a diagnosis of invasive aspergillosis/detection of Aspergillus spp. by culture from sputum, TA, BA, or BALF or positive GM from serum or BALF at time of screening or randomization.
* History of invasive aspergillosis within the prior six months.
* Patients with a known intolerance or hypersensitivity to isavuconazole or other azole agents.
* History of familial short QT syndrome.
* Patients that are being treated with mold-active antifungal agents for invasive aspergillosis or another invasive fungal infection.
* Patients with severe hepatic impairment or liver cirrhosis (Child C) should be excluded from the study unless the treating physicians feel the benefits of treatment outweigh the risks.
* Treatment with Lopinavir/ritonavir for HIV infection.
* Prohibited Medications
* Co-administration with a strong CYP3A4 inhibitor or high-dose ritonavir as they may alter the plasma concentration of isavuconazole.
* Co-administration with a strong CYP3A4 inducer such as rifampin, carbamazepine, St. John's wort, or long acting barbiturates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
The incidence of SARS-CoV-2-associated invasive aspergillosis at time of ICU discharge | From date of admission in ICU assessed up to ICU discharge, approximately 28 days
  A patient with SARS-CoV-2-associated invasive aspergillosis is defined as a patient having COVID-19 infection needing intensive care, mycological evidence of Aspergillus and compatible radiological abnormalities consistent with pulmonary aspergillosis

SECONDARY OUTCOMES:
The incidence of SARS-CoV-2-associated non-Aspergillus invasive fungal infections at time of ICU discharge | From date of admission in ICU assessed up to ICU discharge, approximately 28 days
  A patient with SARS-CoV-2-associated non-Aspergillus invasive fungal infection is defined as a patient having COVID-19 infection needing intensive care, mycological evidence of a non-Aspergillus invasive fungal infection, and compatible radiological abnormalities consistent with non-Aspergillus invasive fungal infection
Survival | From date of admission in ICU assessed up to ICU discharge, approximately 28 days
  Compare the rates of survival at time of discharge from the ICU in those who receive isavuconazole compared to those who receive placebo
Length of ICU stay | From date of admission in ICU assessed up to ICU discharge, approximately 28 days
  Compare the length of ICU stay in those who receive isavuconazole compared to those who receive placebo
Length of Hospital stay | From date of admission in ICU assessed up to hospital discharge, approximately 32 days
  Compare the length of hospital stay in those who receive isavuconazole compared to those who receive placebo
Mortality | At 30 and 90 days
  Compare the mortality rate at 30 and 90 days in those who receive isavuconazole compared to those who receive placebo
Adverse events | From date of start of isavuconazole or placebo through duration of isavuconazole or placebo, approximately 28 days
  Compare the rates of adverse events in those who receive isavuconazole compared to those who receive placebo

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jenks, MD, MPH, Principal Investigator — University of California, San Diego; George Thompson, MD, Study Chair — University of California, Davis; Martin Hoenigl, MD, Study Chair — University of California, San Diego
Locations (3):
- United States (3):
  - University of California Irvine, Orange, California
  - University of California Davis, Sacramento, California
  - University of California San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Permpalung N, Chiang TP, Manothummetha K, Ostrander D, Datta K, Segev DL, Durand CM, Mostafa HH, Zhang SX, Massie AB, Marr KA, Avery RK. Invasive Fungal Infections in Inpatient Solid Organ Transplant Recipients With COVID-19: A Multicenter Retrospective Cohort. Transplantation. 2024 Jul 1;108(7):1613-1622. doi: 10.1097/TP.0000000000004947. Epub 2024 Jun 20. PMID 38419156